CLINICAL TRIAL: NCT01192906
Title: A Phase III, Multi-center, Randomized, 24 Week, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate Efficacy and Safety of RO4917838 in Stable Patients With Persistent, Predominant Negative Symptoms of Schizophrenia Treated With Antipsychotics Followed by a 28 Week, Double-blind Treatment Period.
Brief Title: A Study of RO4917838 (Bitopertin) in Patients With Persistent, Predominant Negative Symptoms of Schizophrenia (WN25309)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN25309; 2010-020467-21
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- 2 (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral doses, once a day for 52 weeks
  Arms: 3
Drug: bitopertin [RO4917838] — Oral dose level 1, once a day for 52 weeks
  Arms: 1
Drug: bitopertin [RO4917838] — Oral dose level 2, once a day for 52 weeks
  Arms: 2

SUMMARY:
This multi-center, randomized, double blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4917838 (bitopertin) in patients with persistent, predominant negative symptoms of schizophrenia. Patients, on stable treatment with antipsychotics, will be randomized to receive daily oral doses of RO4917838 or matching placebo for 52 weeks, followed by an optional treatment extension for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged 18 years and above
* Diagnosis of schizophrenia of paranoid, disorganized, residual, undifferentiated or catatonic subtype
* Predominant negative symptoms
* With the exception of clozapine, patients are on any of the available marketed atypical or typical antipsychotics (treatment with a maximum of two antipsychotics)

Exclusion Criteria:

* Evidence that patient has clinically significant, uncontrolled and unstable disorder (e.g. cardiovascular, renal, hepatic disorder)
* Body Mass Index (BMI) of <17 or >40 kg/m2
* Depressive symptoms, defined as a score of 9 or greater on the Calgary Depression Rating Scale for Schizophrenia (CDSS)
* A severity score of 3 or greater on the Parkinsonism item of the ESRS-A (Clinical Global Impression, Parkinsonism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy (PANSS negative symptoms factor score) | Week 24
Safety (incidence of adverse events) | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (91):
- United States (20):
  - Carson, California
  - Oceanside, California
  - San Diego, California
  - Hartford, Connecticut
  - Norwalk, Connecticut
  - North Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - St Louis, Missouri
  - Omahac, Nebraska
  - Cedarhurst, New York
  - Jamaica, New York
  - Rochester, New York
  - Allentown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
- Brazil (8):
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Pelotas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (10):
  - Calgary, Alberta
  - Medicine Hat, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Montreal, Quebec
  - Verdun, Quebec
- Chile (3):
  - San Miguel
  - Santiago
  - Valdivia
- Germany (7):
  - Berlin
  - Bochum
  - Cologne
  - Freiburg im Breisgau
  - Hamburg
  - München
  - Nuremberg
- Latvia (3):
  - Daugovpils
  - Jelgava
  - Liepāja
- Lithuania (3):
  - Kaunas
  - Šilutė
  - Vilnius
- Netherlands (2):
  - Assen
  - Groningen
- Poland (7):
  - Choroszcz
  - Kielce
  - Lublin
  - Piekary Śląskie
  - Skorzewo
  - Tuszyn
  - Warsaw
- Slovakia (4):
  - Bojnice
  - Bratislava
  - Rimavská Sobota
  - Svidník
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
  - Zamora, Zamora
- Taiwan (6):
  - Hualian Town
  - Kaohsiung City
  - Taichung
  - Tainan
  - Tainan County
  - Taipei
- Turkey (Türkiye) (5):
  - Ankara
  - Diyarbakır
  - Gaziantep
  - Istanbul
  - Manisa
- Ukraine (8):
  - Dnipropetrovsk
  - Donetsk
  - Glevakha Kyviv Region
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Vinnytsia

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Bugarski-Kirola D, Blaettler T, Arango C, Fleischhacker WW, Garibaldi G, Wang A, Dixon M, Bressan RA, Nasrallah H, Lawrie S, Napieralski J, Ochi-Lohmann T, Reid C, Marder SR. Bitopertin in Negative Symptoms of Schizophrenia-Results From the Phase III FlashLyte and DayLyte Studies. Biol Psychiatry. 2017 Jul 1;82(1):8-16. doi: 10.1016/j.biopsych.2016.11.014. Epub 2016 Dec 15. PMID 28117049